CLINICAL TRIAL: NCT07095426
Title: Interplay Between Metabolic Risk Factors, Body Mass Index, and the Gut/Vascular Response to Supplemental Fiber
Brief Title: Impact of Supplemental Fiber on Gut and Vascular Health Related in Obesity Phenotypes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Principal Investigator, Bryant Keirns, Assistant Professor, Ball State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2025-75
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Syndrome; Healthy Participants; Metabolically Healthy Obesity; Metabolically Abnormal Obesity
Keywords: fiber; vascular health; gut health; inflammation
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Metabolically Benign; Inflammation | interventions — Inulin

STUDY DESIGN:
Intervention Model Description: Single arm, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inulin Supplement (Experimental): Participants will consume 6g of pre-portioned powdered inulin from chicory root daily for one week followed by 12g daily for eight weeks. Participants will fully dissolve it into a habitual cool or room temperature beverage to drink around the same time each day.
  Interventions: Dietary Supplement: inulin

INTERVENTIONS:
Dietary Supplement: inulin — 6g inulin from chicory root per day for one week and 12g inulin per day for eight weeks dissolved into cool or room temperature liquid

SUMMARY:
Based on prior research, the investigators are interested in whether an intervention targeting gut health (supplemental fiber for 9 weeks total) will improve vascular health in individuals with obesity. Additionally, the investigators are interested in if this response differs based on whether individuals with obesity have very few heart disease risk factors or several heart disease risk factors.

DETAILED DESCRIPTION:
The investigators will recruit individuals with obesity (body mass index ≥30 kg/m2) from Ball State University Campus and the surrounding community. Participants will be grouped as "metabolically healthy" (0-1 metabolic syndrome risk factors) or "metabolically unhealthy" (≥2 metabolic syndrome risk factors) Participants will be asked to consume inulin for 9 weeks total. Participants will consume 6g of inulin per day during week 1 as a run-in period. The following 8 weeks participants will consume 12g of inulin per day.

Participants will be asked to report for in-lab assessments/visits before the study begins (baseline), halfway through the intervention which starts following the 1-week run-in period (5 weeks), and at the conclusion of the intervention (9 weeks). At all of these assessments, participants will arrive in the morning (roughly 6-10 AM) having fasted for ~10 hours. We will then collect a blood sample, followed by several vascular measurements including flow-mediated dilation, pulse wave analysis, pulse wave velocity, and an electrocardiogram. Body weight and composition will also be assessed using a bioimpedance scale at each visit. Upon completion of each in-lab visit, participants will be asked to wear an ambulatory blood pressure monitoring device for 24 hours and will complete a 3-day food record. Dual-energy X-ray absorptiometry scans will be used to assess body composition at baseline and final study visits. Participants will provide a stool sample collected at home following baseline and final study visits as an optional procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 18-55 years old.
* Participants BMI is ≥30 kg/m2 - this BMI requirement is due to our research aims.
* Participants have either 0-1 or 2+ of the following risk factors outside of the normal reference ranges: blood pressure, blood sugar, triglycerides, and HDL-cholesterol.
* Participants are not pregnant or expecting to become pregnant (females only). •Participants are not postmenopausal (females only).
* Participants have not been diagnosed with an advanced cardiometabolic condition (e.g., cardiovascular disease, type 2 diabetes).
* Participants have not been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease, diverticulosis/diverticulitis).
* Participants do not regularly take anti-inflammatory drugs (more than 2x week) and are willing to suspend use of these medications for 3 days leading up to in-lab visits.
* Participants do not take weight-loss medications (e.g., Ozempic, Wegovy).
* Participants do not use tobacco products or any illicit drugs.
* Participants have not used antibiotics or probiotics in the last month.
* Participants do not have dietary restrictions prohibiting them from consuming the fiber supplement (e.g., food allergies/intolerance).
* Participants do not have a pacemaker.
* Participants are able to lie on their back (supine position) in the dark for at least 10 minutes (related to vascular measurements).

Exclusion Criteria:

* Participants are not 18-55 years old.
* Participants BMI is not ≥30 kg/m2 - this BMI requirement is due to our research aims.
* Participants do not have either 0-1 or 2+ of the following risk factors outside of the normal reference ranges: blood pressure, blood sugar, triglycerides, and HDL-cholesterol.
* Participants are pregnant or expecting to become pregnant (females only).
* Participants are postmenopausal (females only).
* Participants have been diagnosed with an advanced cardiometabolic condition (e.g., cardiovascular disease, type 2 diabetes).
* Participants have been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease, diverticulosis/diverticulitis). •Participants regularly take anti-inflammatory drugs (more than 2x week) and are not willing to suspend use of these medications for 3 days leading up to in-lab visits.
* Participants take weight-loss medications (e.g., Ozempic, Wegovy).
* Participants use tobacco products or any illicit drugs.
* Participants have used antibiotics or probiotics in the last month.
* Participants have dietary restrictions prohibiting them from consuming the fiber supplement (e.g., food allergies/intolerance).
* Participants have a pacemaker.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Serum Soluble Cluster of Differentiation 14 (sCD14) | Through study completion, up to 1.5 years.
  The investigators will measure fasting sCD14 at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Serum Lipopolysaccharide Binding Protein (LBP) | Through study completion, up to 1.5 years.
  The investigators will measure fasting LBP at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Serum C-Reactive Protein (CRP) | Through study completion, up to 1.5 years.
  The investigators will measure fasting CRP at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Heart Rate Variability (HRV) | Through study completion, up to 1.5 years.
  The investigators will measure HRV at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Flow-Mediated Dilation (FMD) | Through study completion, up to 1.5 years.
  The investigators will measure FMD at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Pulse Wave Velocity (PWV) | Through study completion, up to 1.5 years.
  The investigators will measure PWV at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Aortic Aumentation | Through study completion, up to 1.5 years.
  The investigators will measure aortic augmentation at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Augmentation Index (AIx) | Through study completion, up to 1.5 years.
  The investigators will measure AIx at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.

SECONDARY OUTCOMES:
Blood Pressure | Through study completion, up to 1.5 years.
  The investigators will measure peripheral, central, and ambulatory blood pressure at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Glucose | Through study completion, up to 1.5 years.
  The investigators will measure fasting glucose at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
High-Density Lipoprotein Cholesterol (HDL-C) | Through study completion, up to 1.5 years.
  The investigators will measure fasting HDL-C at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Triglycerides | Through study completion, up to 1.5 years.
  The investigators will measure fasting triglycerides at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Digestive Symptoms | Through study completion, up to 1.5 years.
  The investigators will measure digestive symptoms at each visit. These measurements will take place immediately and a complete dataset will be compiled upon study completion.

OTHER OUTCOMES:
Body Composition | Through study completion, up to 1.5 years.
  The investigators will measure body composition using bioelectrical impedance and waist circumference at each visit, and dual-energy X-ray absorptiometry at the baseline and final visits. These measurements will take place immediately and a complete dataset will be compiled upon study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Keirns, PhD, Principal Investigator — Ball State University
Locations (1):
- Health Professions Building, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided